CLINICAL TRIAL: NCT05411419
Title: Spinal Cord Stimulation for the Management of Chronic Non-cancer Pain: a Retrospective Study
Brief Title: Retrospective Analysis of Spinal Cord Stimulation on Chronic Non-cancer Pain
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chi-Wai Cheung, Professor, The University of Hong Kong
Other Study IDs: UW22-507
Record Dates: First submitted 2022-06-05; First posted 2022-06-09 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spinal cord stimulation — Two leads for spinal cord stimulation would be implanted.

SUMMARY:
Since 2014, the Queen Mary Hospital, a tertiary teaching hospital in Hong Kong, has commenced the provision of spinal cord stimulation (SCS) services with structured guidelines, standardized protocols and comprehensive pre- and post-operative assessments. It is hoped that the needs of chronic pain patients, especially those who are refractory to conventional medical management, can be better addressed with the introduction of SCS. Hence, through the proposed retrospective study, the investigator aim to systematically evaluate the use of SCS in Queen Mary Hospital, thereby providing evidence with regard to its efficacy and safety for pain management.

DETAILED DESCRIPTION:
As one of the most common health complaints in the world, low back pain (LBP) can affect people across all age groups, with a lifetime prevalence of 84%. In Hong Kong LBP is reported to be the second most prevalent illness due to work and the most common illness made worse by work. LBP can be acute or chronic, with the former lasting less than six weeks and the latter lasting more than twelve weeks. LBP is believed to have an adverse impact on quality of life and functional performance, creating social and economic costs.

Current guidelines on the management of chronic LBP generally recommend the use of conservative treatments, pharmacological agents and/or invasive treatments. Non-steroidal anti-inflammatory drugs (NSAIDs) are commonly used in pharmacologic therapy, while conservative treatments such as supervised exercise therapy and cognitive behavioural therapy are other possible therapeutic options. If necessary, more invasive treatments including epidural corticosteroids, intra-articular steroid injections and spinal cord stimulation may be considered.

With the advances in neuromodulation in recent decades, spinal cord stimulation (SCS) has become a well-established therapeutic modality for the treatment of chronic pain. Through the delivery of electrical stimulation to the dorsal column of the spinal cord, SCS modulates the pain signals and replaces the pain sensation with tingling paraesthesia for pain relief. Evidence-based guidelines published by the Neuromodulation Appropriateness Consensus Committee (NACC) of the International Neuromodulation Society recommend the use of SCS for a variety of chronic pain conditions, which include failed back surgery syndrome (FBSS), complex regional pain syndrome (CRPS), upper extremity neuropathic pain syndrome, chronic refractory angina and ischemic peripheral neuropathic pain.

Yet the effectiveness of SCS on chronic non-cancer pain management is still unknown in Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* all patients underwent SCS for chronic non-cancer pain management between 2014 to 2021 in Queen Mary Hospital

Exclusion Criteria:

* missing of essential data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data of all patients underwent SCS between 2014 to 2021 for non-cancer pain management kept in the Pain Clinic, Queen Mary Hospital would be retrieved.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
pain score | At 1 week after implant of spinal cord stimulation
  Pain score using numerical rating scale (NRS) from 0 to 10, 0 represents no pain, and 10 represents the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No